CLINICAL TRIAL: NCT00118690
Title: A Stratified, Multicenter, Randomized, Double-Blind, Parallel Group, 4-Week Comparison of Fluticasone Propionate/Salmeterol DISKUS Combination Product 100/50mcg BID Versus Fluticasone Propionate DISKUS 100mcg BID in Pediatric and Adolescent Subjects With Activity-Induced Bronchospasm
Brief Title: A Study Measuring Asthma Control In Pediatric And Adolescent Subjects Whose Asthma Is Worsened By Activity Or Exercise
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SFA100316
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Bronchospasm; Activity/Exercise Induced Bronchospasm
Keywords: bronchospasm; asthma
MeSH Terms: conditions — Bronchial Spasm; Motor Activity; Asthma, Exercise-Induced; Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fluticasone propionate/salmeterol

SUMMARY:
During this study, your child will need to attend up to 5 office visits and maintain regular telephone contact with the clinic. Certain office visits will include physical exams, medical history review, exercise challenge test (walking/running on a treadmill), electrocardiogram (ECG) tests, and lung function tests. All study related medications and medical examinations are provided at no cost. All study drugs are currently available by prescription to patients 4 years and older.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with persistent asthma for 3 months or longer.
* Experience worsened asthma symptoms during physical activity.
* Using or used an inhaled steroid for the last 4 weeks or longer (such as Aerobid, Azmacort, Flovent, Pulmicort, QVAR, or Vanceril).

Exclusion criteria:

* Used systemic steroids as either liquids, pills, or injections to treat asthma within the last 3 months.
* Have only intermittent, seasonal, or exercise induced asthma, and not persistent asthma.
* Admitted to a hospital within the last 6 months due to asthma symptoms.
* Any poorly controlled medical conditions that may make study participation unsafe or inappropriate in the opinion of the study physician (such as cystic fibrosis, congenital heart disease, insulin dependent diabetes, glaucoma, drug allergies, etc.).
* The study physician will evaluate other medical criteria.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 227 (Actual)
Dates: Start 2003-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in maximal decline from baseline in lung function following exercise challenge after 4-weeks of double-blind treatment compared to decline in lung function before treatment.

SECONDARY OUTCOMES:
Daily lung function tests and subject assessed diary measures analyzed over the 4-week treatment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (48):
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, East Artesia, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Madera, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Rolling Hills Est, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Pueblo, Colorado
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Robbinsdale, Minnesota
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Mount Laurel, New Jersey
  - GSK Investigational Site, Kernersville, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: http://www.findclinicalstudy.com — http://www.findclinicalstudy.com
- Available data/document: Clinical Study Report: SFA100316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SFA100316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SFA100316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SFA100316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SFA100316 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register